CLINICAL TRIAL: NCT05137470
Title: Study on the Changes of Emotion and Cognitive Function and Brain Imaging in Uremic Patients Before and After Entering Dialysis
Brief Title: Emotion and Cognitive Function and Brain Imaging Change in HD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YYYXYJ-2021-275
Record Dates: First submitted 2021-11-24; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-10

CONDITIONS: Kidney Failure, Chronic; Cognitive Dysfunction; Magnetic Resonance Imaging
MeSH Terms: conditions — Kidney Failure, Chronic; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly HD patients: Newly admitted patients with uremia who started hemodialysis treatment
  Interventions: Other: This is an observational study
- MHD patients: Maintenance hemodialysis patients
  Interventions: Other: This is an observational study

INTERVENTIONS:
Other: This is an observational study — This is an observational study

SUMMARY:
1. Observe the influence of entering hemodialysis treatment on the emotional and cognitive functions of ESRD patients.
2. Observe the influence of entering hemodialysis treatment on the brain structure imaging of ESRD patients.
3. Analyze and study the relevant clinical risk factors of the above-mentioned effects, and find targets for therapeutic intervention.

DETAILED DESCRIPTION:
Select uremic patients and maintenance hemodialysis patients admitted to the Central Dialysis Room of Beijing Friendship Hospital, Capital Medical University from 2021, to collect and sort out the demographic characteristics of the patients: gender, age, clinical characteristics: primary disease, complications and Complications, body mass index (BMI), residual renal function, etc., clinical examination indicators: hemoglobin, blood calcium, blood phosphorus, blood PTH, blood albumin, URR, etc., hemodialysis treatment parameters: dialysis mode, dialyzer model, vascular access , Blood flow, etc., record the patient's emotional and cognitive function status, various clinical indicators and changes in the patient's quality of life before and after the start of treatment, and use multimodal magnetic resonance neuroimaging research sequences to analyze the changes in the patient's brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are new to hemodialysis treatment, and those who are on regular hemodialysis treatment for ≥6 months.
* Age ≥ 18 years old.

Exclusion Criteria:

* There was already a severe central nervous system disease before dialysis.
* Hearing and visual impairment cannot communicate or cooperate.
* Mental illness and incapacity.
* The magnetic resonance examination could not be completed for various reasons.
* Life expectancy with serious diseases is less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Uremia patients undergoing hemodialysis treatment in the hemodialysis room of Beijing Friendship Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Appears obvious emotional and cognitive decline, or abnormal head MRI | 2 years
  Appears obvious emotional and cognitive decline, or abnormal head MRI

CONTACTS AND LOCATIONS:
Overall Officials: WENHU LIU, doctor, Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No